CLINICAL TRIAL: NCT02314416
Title: Stem Cells In Wound Healing With Collagen Matrix as a Carrier
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: NuTech Medical, Inc (Industry)
Responsible Party: Principal Investigator, Edmond Ritter, Professor of Plastic and Reconstructive Surgery, Augusta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 611757
Record Dates: First submitted 2014-12-08; First posted 2014-12-11 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Wounds
Keywords: wounds, stem cells, collagen matrix, maturation
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Treatment (Active Comparator): Patients in the Control Arm will receive collagen matrix for wound coverage and standard wound care that will include chemical/surgical debridement (using a topical paste to clean the wound or removing bad tissue using a scalpel or scissors) and dressing care. In addition, they may also have imaging studies (such as x-ray, CAT scan, ultrasound) performed if determined to be necessary by the physician.
  Interventions: Biological: Amniotic Stem Cells and Collagen Matrix
- Amniotic Stem Cells and Collagen Matrix (Experimental): Patients will receive amniotic stem cells(NuCel) embedded in collagen matrix for wound coverage, and standard wound care that will include chemical/surgical debridement (using a topical paste to clean the wound or removing bad tissue using a scalpel or scissors) and dressing care. In addition, they may also have imaging studies (such as x-ray, CAT scan, ultrasound) performed if determined to be necessary by the physician.
  Interventions: Biological: Amniotic Stem Cells and Collagen Matrix

INTERVENTIONS:
Biological: Amniotic Stem Cells and Collagen Matrix — Nucel will be applied in between two pieces of collagen matrix'. The NuCel-impregnated collagen matrix will be placed over a clean, debrided wound.
  Other Names: NuCel

SUMMARY:
The purpose of the study is to use a collagen matrix embedded with amniotic stem cells to speed up the maturation and integration of the collagen matrix in the wound bed and shorten total time needed for wound healing.

DETAILED DESCRIPTION:
Wounds are a widespread problem all around the world. From a practical purpose, wounds are divided in acute and chronic. Acute wound management depends on amount and type of tissue destruction. Therefore, acute wounds could be furthermore subdivided as simple wound where only skin is missing and complex wounds when some underlying structures are involved. Complex wounds may require free flap if wound beds are poorly vascularized, devascularized or underlying tissue wouldn't accept skin graft or biologically derived extracellular matrix (BDEM). Simple wounds, on other hand, would be managed in the past by skin graft or by local flap when feasible. These management strategies commonly result in unacceptable aesthetically and/or functionally (e.g. contracture, unstable wound) outcomes and will often require secondary reconstruction.

The second class of wounds is the chronic wounds. Chronic wounds occur whenever the normally well-orchestrated reparative process does not proceed in a sequential and timely fashion from hemostasis and inflammation, through proliferation to remodeling. The process is necessarily complicated and can be delayed by many intrinsic and extrinsic factors along the way (1). Acute and chronic wounds pose a significant burden to patients, healthcare professionals, and the healthcare system, affecting more than 15.5 million patients and costing an estimated $ 500 billion annually (2-3). Based on their pathogenesis, there are four principle types of chronic wounds: venous ulcers, diabetic ulcers, arterial ischemic and pressure ulcers.

1. Venous ulcers usually occur in the legs, account for the majority of wounds, and often affecting the elderly with prior history of deep venous thrombosis (DVT). Ulcers form eventually, when cells cannot keep with rate of degradation.
2. Diabetic ulcers are seen in diabetic patients who are developing ulcers for several reasons. Neuropathy and micro-angiopathy are quite common, and these changes together with a reduced immunity set up the perfect storm for tissue breakdown in the lower extremities. Because of all these factors, exacerbated by impaired healing, even the smallest cuts or bruises can become dangerously infected.
3. PAD, is a term that covers an array of medical problems caused by obstruction of the large arteries in the arms or legs. In the advanced form of PAD, critical limb ischemia (CLI) can occur, which is a leading cause of lower limb amputations. The Angiogenesis Foundation estimates that 1.4 million people in the United States have CLI, with an estimated 350,876 new cases diagnosed each year (2).
4. Pressure ulcers comprise the fourth major type of wounds. These typically occur in people who are bedridden or whose mobility is severely limited. They are caused by a loss of blood circulation that occurs when pressure on the tissue is greater than the perfusion pressure in capillaries, thereby cutting off circulation, rendering tissue ischemic. The combination of anesthesia and paralysis is a potent inducer of tissue break down. Data from spinal cord units at Veterans Affairs Medical Centers show an alarmingly high prevalence and incidence of pressure ulcers in young soldiers paralyzed by spinal cord injuries.

Over the past decades, little improvement has been made in reducing morbidity and disability from chronic wounds (3). The best available treatment for chronic wounds achieves only a 50% healing rate that is often temporary, with an unacceptably high recurrence rate. Among the many factors contributing to "stalling" of wound healing processes, impairment in the production of cytokines by local inflammatory cells and fibroblasts and reduced angiogenesis are crucial problems (4).

The introduction of BDEMs has improved wound care significantly over the years. The most commonly used BDEM is a bovine derived collagen matrix. This bovine collagen matrix is a FDA approved wound care device comprised of a porous matrix of cross-linked bovine tendon collagen and glycosaminoglycan and a semi-permeable polysiloxane (silicone layer). The collagen-glycosaminoglycan biodegradable matrix provides a scaffold for cellular invasion and capillary growth (5). The use of the bovine collagen matrix can improve aesthetic and functional outcomes in complex wounds with full thickness skin defects and exposure of underlying structure such as muscle, tendons, vessels or nerves. Despite its clinical benefit, a significant problem exists due to the long period required for vascularization and regeneration, which requires 3 weeks as per the manufacturer. As a result, this not only increases the cost of wound management but also decreases income potential and quality of life.

As research is being advanced in the field of wound care, stem cell therapy is emerging to be a promising approach to the treatment of both acute and chronic wounds. It is now known that bone marrow-derived stem cells (BMSC) are multipotential stem cells capable of differentiation into numerous cell types including fibroblast, muscle, brain, and cartilage (6). Among the cells found in BMSCs is a group called mesenchymal stem cells (MSC). MSCs are stromal cells that have been held in reserve with the ability to self-renew and also exhibit multilineage differentiation. MSCs are also found in fetal and adult tissues and have been isolated from umbilical cord, endometrial polyps, adipose tissue, and menstrual blood. Because they are readily available to harvest from various tissues, MSCs are an attractive choice in experimental and possible clinical applications.

Recent clinical observations and small sample size studies report accelerated healing in difficult wounds by topical and regional applications of mononuclear cell preparations from autologous bone marrow. In the rat model, the application of systemic and local BMSCs have has resulted in improved wound healing through increased wound tensile strength, increased collagen, and faster wound maturation (7). However, bone marrow harvesting is painful, at times requires general anesthesia, and occasionally not feasible due to the debilitated state of the patients. It is thus, extremely desirable to use off-the-shelf, commercially available, allogeneic, mesenchymal stem cells.

NuCel (NutechMedical, Birmingham, AL USA) is a FDA approved allograft containing MSCs derived from human amnion and amniotic fluid and is currently being used in different clinical settings including orthopedic surgery and in neurosurgery as grafts. Amnion-derived MSCs have been reported to have high trans-differentiation and angio-vasculogenic properties (8). NuCel stem cells are immune privileged as the do not express major histo-compatibility complex class II and has lower expression of MHC class I compared with adult bone marrow derived stem cells. NuCel contains five types of collagen and fibronectin which are factors involved in the wound healing process. Moreover, they are less ethically controversial due to the abundance of waste placenta.

Multiple studies have shown that pluripotent stem cells can increase and speed up vascularization of BDEM and significantly decrease the time to BDEM maturation (6-8). As a result, there is potential for this application to decrease the cost of wound management and increase quality of life.

In summary, we propose to test definitively, the safety and effectiveness of just such allogeneic MSCs, NuCel, in promoting the healing of acute and chronic wounds. NuCel consists of a special class of human stem cells that have the ability to express a range of therapeutically relevant proteins and other factors, as well as form multiple cell types. We propose a pilot study is to be conducted at the Georgia Regents University. It is a prospective, randomized, controlled trial with the aim to generate Level I and II evidence on the effectiveness of amniotic stem cells using a collagen matrix as a carrier in enhancing healing of wounds.

The goal and design of the current proposal is to establish a practical protocol which has the potential to not only accelerate the translation of advances in knowledge into new standards of care for wound management, but also is safe, FDA approved, and inexpensively accessible to address some of the most pressing needs in today's wound healing field. The main objective of the current proposal is to use amniotic MSC to speed up maturation and integration of collagen matrix in the wound bed and shorten total time needed for wound healing. This can potentially result in a saving of hundreds of millions of dollars to the healthcare system. The outcome of this proposal will accelerate translation of greater medical capabilities to patients using a novel, safe and creative intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an acute or chronic would that present for a plastic surgery consultation for wound care.

Exclusion Criteria:

* Active Smokers,
* Immunosuppressed patients,
* nutritionally depleted patients,
* terminally ill cancer patients,
* transplant patients,
* ASA class IV and higher will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Maturation of Collagen Matrix (Changes in color of collagen matrix from tan to white to vanilla, which signifies vascularity) | Days 3, 5, 7, 14, 21 and 28 after treatment
  Changes in color of Collagen Matrix from tan to white to vanilla, which signifies vascularity

SECONDARY OUTCOMES:
Complete Wound Healing (Change is size of wound in millimeters) | Days 3, 4, 7, 14, 21 and 28 after treatment
  Change is size of wound in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Edmond Ritter, MD, Principal Investigator — Professor of Plastic Surgery and Reconstructive Surgery